CLINICAL TRIAL: NCT00113906
Title: The Effect of Melatonin Treatment on Postoperative Fatigue and Sleep Disturbances: A Placebo Controlled Randomized Clinical Trial
Brief Title: Melatonin Treatment After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-003796-37
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2005-06

CONDITIONS: Postoperative Complications; Fatigue; Dyssomnias
Keywords: melatonin,; fatigue,; sleep quality,; circadian,; postoperative; Postoperative fatigue; postoperative sleep disturbance; general wellbeing
MeSH Terms: conditions — Postoperative Complications; Fatigue; Dyssomnias; Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: melatonin

SUMMARY:
Circadian disturbances occur after surgery. A double blinded, placebo controlled randomized clinical trial was made to investigate effects of melatonin on postoperative fatigue, sleep disturbances and general wellbeing.

DETAILED DESCRIPTION:
Postoperative fatigue and sleep disturbances occur after minimally invasive surgery. The pathophysiological background is unknown, but several studies have shown disturbed melatonin secretion after surgery. It is unknown whether melatonin substitution will improve general wellbeing, fatigue or sleep disturbances after laparoscopic cholecystectomy. We set out to study in a randomized clinical trial to investigate the effect of 5 mg melatonin versus placebo, on postoperative sleep disturbances, fatigue and general wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Operation for gall bladder disease
* Age over 18 years

Exclusion Criteria:

* Known preoperative sleep disturbance
* Anticoagulant therapy
* Psychiatric disease
* Lack of written informed consent
* Treatment with hypnotics within one week prior to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Fatigue

SECONDARY OUTCOMES:
Sleep quality
general wellbeing
pain

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, MD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (2):
- Denmark (2):
  - University Hospital of Glostrup, Glostrup Municipality, Copenhagen
  - Copenhagen University Hospital, Gentofte, Hellerup, Copenhagen